CLINICAL TRIAL: NCT00353899
Title: Cardiovascular Magnetic Resonance Imaging of Pediatric Healthy Volunteers
Brief Title: Cardiovascular Magnetic Resonance Imaging of Pediatric Normal Volunteers
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060208; 06-H-0208
Record Dates: First submitted 2006-07-18; First posted 2006-07-19 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2017-04-26

CONDITIONS: Healthy
Keywords: Magnetic Resonance Imaging; Pediatric; Normal Volunteer; Electrocardiogram; Cardiac; Healthy Volunteer; HV

SUMMARY:
This study will examine ways to establish and standardize normal measurements for children, specific to gender, age, and body surface, when using magnetic resonance imaging (MRI). MRI, which was introduced in the 1980s, is being used more frequently for children. In this study, researchers seek to understand how a child's heart is different from that of an adult, when an MRI is used for tests. More children with congenital heart disease are living longer. Researchers are looking for a better way to assess their cardiac anatomy and function, and to compare findings with normal function.

Patients ages 8 to 21 in good health and who do not smoke may be eligible for this study. There will be a blood or urine test to check for pregnancy in female volunteers who have begun menstruating or who are over age 12. Pregnancy test results must be negative for those patients to stay in the study. The MRI technique uses a strong magnetic field and radio waves to obtain images of body organs and tissues. For that procedure, patients will lie still on a table that slides into the enclosed tunnel of the scanner. They will be in the scanner from 20 to 60 minutes. As the scanner takes pictures, patients will hear knocking or beeping sounds, and they will wear earplugs to reduce the noise. Patients will be able to communicate with the MRI staff at all times during the scan. At any time, patients or their parents may ask that the patients be moved out of the machine. If they would like, patients can bring a music CD or listen to a radio station through headphones. Some MRI techniques require monitoring while the patient is undergoing the scan. For monitoring of the heart, an electrocardiogram (EKG) will be performed to make sure that the heart rhythm is normal and that heart disease is not present. Patients may be asked to wear adhesive patches that are attached to wires of the EKG machine on their chests. To monitor breathing, patients may be asked to wear a rubber belt that stretches as they take a breath. So that the best quality images are produced, patients may be asked to hold their breath for about 15 seconds.

During the MRI scan, patients may experience peripheral nerve stimulation, usually experienced as a muscle twitch. It is caused by rapid switching of magnetic fields and is not serious. Patients who feel a muscle twitch should report that sensation to the person performing the scan. It is possible, though unlikely, for a painful sensation to result from nerve stimulation. Patients should immediately report if they have pain so that the scan can be stopped.

DETAILED DESCRIPTION:
A cardiac MRI (Magnetic Resonance Imaging) scan will be performed on normal children and young adult volunteers. These studies will be conducted in the MRI systems located in the NIH Clinical Center in Bethesda, Maryland. The results will be used to establish the normal standard MRI measurements for the pediatric population; including left ventricular mass, ejection fractions and other standard cardiac measurements.

ELIGIBILITY:
* INCLUSION CRITERIA:

Any normal volunteer between the ages of 8 and 21 years old, non-smoker who is capable of giving assent and has a legal guardian to give informed consent if under 18 years old.

EXCLUSION CRITERIA:

A subject will be excluded if he/she has a contraindication to MR scanning.

1. Brain aneurysm clip
2. Implanted neural stimulator
3. Implanted cardiac pacemaker or defibrillator
4. Cochlear implant
5. Ocular foreign body (e.g. metal shavings)
6. Insulin pump

<TAB>

To assess whether subjects are indeed normal, the legal guardian will be asked to fill out a questionnaire. Subjects also will be excluded for a paralyzed hemidiaphragm, morbid obesity (BMI greater than 30%), claustrophobia, smokers, significant asthma (greater than one asthma attack per month for the past three months), pregnancy, major medical illness requiring regular medications (such as steroids that may alter muscle mass, sickle cell disease, thalassemia), history of cardiac disease (requiring SBE prophylaxis when visiting the dentist), and/or history of significant previous surgery that may alter cardiac anatomy (such as diaphragmatic hernia, tracheoesophageal fistula).

Females of menstruating age will receive a pregnancy test as part of the screening process to participate in this protocol. If they do not wish to be tested, they cannot participate in this voluntary protocol.

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2006-07-14; Study Completion 2017-04-26

CONTACTS AND LOCATIONS:
Overall Officials: Andrew E Arai, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Sierra-Galan LM, Ingkanisorn WP, Rhoads KL, Agyeman KO, Arai AE. Qualitative assessment of regional left ventricular function can predict MRI or radionuclide ejection fraction: an objective alternative to eyeball estimates. J Cardiovasc Magn Reson. 2003 Jul;5(3):451-63. doi: 10.1081/jcmr-120022261. PMID 12882076
- [Background] Lorenz CH. The range of normal values of cardiovascular structures in infants, children, and adolescents measured by magnetic resonance imaging. Pediatr Cardiol. 2000 Jan-Feb;21(1):37-46. doi: 10.1007/s002469910006. PMID 10672613
- [Background] Lorenz CH, Walker ES, Morgan VL, Klein SS, Graham TP Jr. Normal human right and left ventricular mass, systolic function, and gender differences by cine magnetic resonance imaging. J Cardiovasc Magn Reson. 1999;1(1):7-21. doi: 10.3109/10976649909080829. PMID 11550343